CLINICAL TRIAL: NCT02898844
Title: Randomized Controlled Experiment of Dieting in Pairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A. Janet Tomiyama (Other)
Responsible Party: Sponsor-Investigator, A. Janet Tomiyama, Faculty Sponsor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-000666
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Dietary Modification
Keywords: dieting; dyads; psychological well-being; weight loss; cortisol
MeSH Terms: conditions — Psychological Well-Being; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Condition (No Intervention): Neither roommate dieted.
- Mixed Diet Condition (Experimental): Low-calorie diet: One roommate in each pair was randomly assigned to a 1200-calorie/day diet, while the other roommate was instructed to eat normally.
  Interventions: Behavioral: Mixed Diet Condition
- Both Diet Condition (Experimental): Low-calorie diet: Both roommates in each pair were randomly assigned to a 1200-calorie/day diet.
  Interventions: Behavioral: Both Diet Condition

INTERVENTIONS:
Behavioral: Mixed Diet Condition — One roommate dieted and the other ate normally.
  Arms: Mixed Diet Condition
Behavioral: Both Diet Condition — Both roommates dieted.
  Arms: Both Diet Condition

SUMMARY:
This study examined how dieting with a partner affects weight loss, diet adherence, psychological well-being, and cortisol.

DETAILED DESCRIPTION:
The goal of this study was to understand how different types of diet "buddy systems" affect diet success and outcomes related to dieting. Pairs of non-romantic cohabiting female dyads (i.e. roommates) were randomly assigned to one of the following three-week manipulations: (a) neither roommate dieted, (b) one roommate was assigned to a 1200-calorie/day diet and the other ate normally, (c) both roommates were assigned to a 1200-calorie/day diet. Both pre- and post diet, participants were weighted and measured, filled out psychological questionnaires, and provided two days of diurnal salivary cortisol samples. During the three-week manipulation period, participants who were assigned to diet recorded all calories consumed on each day. This study tested whether dieting in a pair would lead to improved diet outcomes in terms of adherence and weight loss, changes in psychological well-being, and changes in cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over 18 years of age
* Interested in dieting in the coming 12 months
* self-reported BMI over 18.5
* < 5 kg weight change in previous 3 months
* Have a university meal plan
* Have a roommate also willing/eligible to participate

Exclusion Criteria:

* Recent/current history of major medical disorder
* Pregnancy/lactation
* History of eating disorder
* Use of lipid-lowering medications
* Use of weight-altering/metabolism-altering medications
* Smoking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Psychological well-being measured via electronic questionnaires | ~3 days after end of 3-week manipulation
Weight loss measured via pounds | ~3 days after end of 3-week manipulation
Diet adherence measured via daily calorie counts | up to 3-week

SECONDARY OUTCOMES:
Cortisol measured via 2 days diurnal cortisol | 1 day after end of 3-week manipulation

CONTACTS AND LOCATIONS:
Overall Officials: A. Janet Tomiyama, PhD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spielberger CD, Gorsuch RL, Lushene RE. State-trait anxiety inventory (self-evaluation questionnaire). Consulting Psychologists Press: 1970.
- [Background] Radloff, L. S. The CES-D scale a self-report depression scale for research in the general population. Applied psychological measurement, 1(3): 385-401, 1977.
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417